CLINICAL TRIAL: NCT07372911
Title: Corneal Wavefront Guided PRK Combined With Epi-off Corneal Cross-Linking Versus Epi-off Corneal Cross-Linking With PTK Epithelial Removal in Keratoconus: A Randomized Clinical Trial
Brief Title: PRoTECT: Corneal Wavefront Guided PRK + Epi-off CXL vs. PTK+Epi-off CXL in Keratoconus
Acronym: PRoTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRoTECT-CXL-TGPRK-MX
Record Dates: First submitted 2025-11-16; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Keratoconus
Keywords: Keratoconus; Corneal ectasia; Corneal cross-linking; Corneal collagen crosslinking (CXL); Epi-off CXL; Riboflavin UV-A; Topography-guided PRK; TG-PRK; Phototherapeutic keratectomy (PTK); PTK epithelial removal; Schwind AMARIS excimer laser; Excimer laser; Athens Protocol (TG-PRK + CXL); Crete protocol (PTK + CXL); Pentacam Scheimpflug tomography; Kmax; Higher-order aberrations (HOAs); Corneal haze; Specular microscopy; Endothelial cell density; NEI VFQ-25; Visual acuity (logMAR); Randomized clinical trial; Parallel assignment
MeSH Terms: conditions — Keratoconus; Corneal Opacity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corneal Wavefront Guided PRK + CXL (Experimental): Corneal wavefront guided therapeutic PRK (50 µm) with Schwind AMARIS, followed by accelerated epi-off CXL. Intensity: 30 mW/cm² (pulsed 1 s on / 1 s off; 50% duty cycle). Total energy (fluence): 5.4 J/cm². Total time (elapsed): 6 minutes [equivalent to 3 minutes "on" time].
  Interventions: Device: Schwind AMARIS excimer laser; Procedure: Corneal collagen crosslinking epi-off accelerated
- PTK + CXL (Active Comparator): Epithelial removal by PTK using Schwind AMARIS, followed by accelerated epi-off CXL. Intensity: 30 mW/cm² (pulsed 1 s on / 1 s off; 50% duty cycle). Total energy (fluence): 5.4 J/cm². Total time (elapsed): 6 minutes [equivalent to 3 minutes "on" time].
  Interventions: Device: Schwind AMARIS excimer laser; Procedure: Corneal collagen crosslinking epi-off accelerated

INTERVENTIONS:
Device: Schwind AMARIS excimer laser — Used for corneal wavefront guided PRK therapeutic ablation (50 µm) or for PTK epithelial removal, according to arm assignment.
Procedure: Corneal collagen crosslinking epi-off accelerated — Riboflavin-UVA crosslinking performed after epithelial removal (corneal wavefront guided PRK arm via PRK; comparator arm via PTK). Intensity: 30 mW/cm² (pulsed 1 s on / 1 s off; 50% duty cycle). Total energy (fluence): 5.4 J/cm². Total time (elapsed): 6 minutes [equivalent to 3 minutes "on" time].

SUMMARY:
Keratoconus causes irregular astigmatism and reduced vision. Epi-off corneal crosslinking (CXL) stabilizes the cornea but often leaves higher-order aberrations uncorrected. This randomized, parallel-group trial compares corneal wavefront guided photorefractive keratectomy (corneal wavefront guided PRK, 50 µm therapeutic ablation) combined with accelerated epi-off CXL versus epi-off CXL with epithelial removal by phototherapeutic keratectomy (PTK) using a Schwind AMARIS excimer laser, in adults with keratoconus. The primary endpoint is change in best-corrected distance visual acuity (logMAR) at 12 months. Key secondary endpoints include Kmax, corneal higher-order aberrations, manifest refraction, Scheimpflug densitometry (haze) and Fantes grade, Corvis ST biomechanics, NEI VFQ-25, and endothelial cell density by non-contact specular microscopy at 1, 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Diagnosis of keratoconus, ABCD Belin stage I-III at baseline
* Minimum (thinnest) corneal pachymetry ≥ 450 µm pre-op
* Written informed consent
* Age-stratified progression requirements:
* 18-25 y: keratoconus stage I-III (progression not mandatory)
* 25-35 y: documented progression (meet ≥ 2 Table-1 criteria below) or, if recent documentation is absent, high-risk features for future progression: Kmax > 53 D, strong family history, severe atopy with persistent eye rubbing, or any of the following over 12 months: ΔKmax ≥ 1.0 D, thinnest pachymetry decrease ≥ 10 µm, or increase in manifest cylinder ≥ 1.0 D
* 35-40 y: clear, unequivocal recent progression (meet ≥ 2 Table-1 criteria); late-onset documented progression may be considered

Exclusion Criteria:

* Central corneal scars or opacities
* Prior ocular surgery or trauma (exception: prior LASIK if it is the cause of post-surgical ectasia, per protocol text)
* Autoimmune disease or uncontrolled diabetes mellitus
* Pregnancy or lactation
* Contact lens wear within 2 weeks before baseline evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in best-corrected distance visual acuity (logMAR) | Baseline to 12 months
  ETDRS-based CDVA in logMAR; change from baseline at 12 months; primary analysis by ANCOVA adjusted for baseline; one study eye per participant.

SECONDARY OUTCOMES:
Change in Kmax (Diopters) | Baseline; 3; 6; 12 months
  Pentacam Scheimpflug tomography; maximum keratometry (D); change from baseline at each time point.
Change in corneal higher-order aberrations (µm RMS) | Baseline; 3,6,12 months
  Wavefront/aberrometry total HOAs RMS (µm) over 6-mm pupil; change from baseline.
Change in manifest refraction spherical equivalent (Diopters) | Baseline; 3;6;12 months
  Manifest refraction SE (D); change from baseline.
Corneal haze (Scheimpflug densitometry units) | Baseline; 3;6;12 months
  CCT and corneal haze as measured by Pentacam Corneal Densitometry. Unit of measure: gray units.
Corvis ST metric: Ambrosio Relational Thickness horizontal (ART-h) | Baseline; 3,6; 12 months
  ART-h as measured by Corvis ST. Unit of measure: microns
Visual Functioning Questionnaire (NEI VFQ-25) | Baseline; 6;12 months
  NEI VFQ-25 composite and subscale scores computed per scoring manual; change from baseline. 0 to 100, where higher scores indicate better vision-related quality of life.
Endothelial cell density (cells/mm²; specular microscopy) | Baseline; 1; 3; 6; 12 months
  Non-contact specular microscopy; primary metric = endothelial cell density (cells/mm²); secondary metrics (if collected) = coefficient of variation and hexagonality; change from baseline; one study eye per participant.
Serious corneal adverse events | Baseline to 12 months
  Incidence of protocol-defined serious ocular AEs ( infectious keratitis, perforation, persistent epithelial defect >14 days, ≥20% endothelial cell density loss, visually significant stromal scarring requiring surgery).
Corneal haze (Fantes grade) | Baseline; 3; 6; 12 months
  Fantes clinical haze grade (ordinal); recorded at each visit. Units: Fantes grade. Scale: 0-4 scale, higher scores = worse haze.
Corvis ST metric: Inverse Concavity Radius | Baseline; 3; 6; 12 months
  Inverse Concavity Radius as measured by Corvis ST. Unit of measure: mm

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmología FAP Conde de Valenciana, IAP Sede Centro, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided